CLINICAL TRIAL: NCT02381093
Title: Does Contextual Interference Improve Retention of Basic Life Support Skills? A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: OttawaHRI
Record Dates: First submitted 2015-03-02; First posted 2015-03-06 (Estimated); Last update posted 2017-12-19 (Actual); Status verified 2017-12

CONDITIONS: Basic Life Saving Skills; Cardiopulmonary Resuscitation; Skill Retention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard BLS Course (Active Comparator): Participants will partake in a standard BLS course.
  Interventions: Other: Standard BLS Course
- Contextual Interference (Experimental): Participants will partake in a BLS course designed using contextual interference scheduling.
  Interventions: Other: Modified BLS course

INTERVENTIONS:
Other: Modified BLS course — BLS using CI
  Arms: Contextual Interference
Other: Standard BLS Course — Usual BLS teaching
  Arms: Standard BLS Course

SUMMARY:
The current method of teaching Basic Life Support (BLS) courses involves a practice schedule where learners rotate through each station once, without repetition. Laypeople learning within this blocked schedule may experience poor skill retention, resulting in suboptimal delivery of Cardiopulmonary Resuscitation (CPR). Implementing a Contextual Interference (CI) practice scheduling method to BLS training would involve presenting each station multiple times within the same timeframe. CI is known to lead to better retention in other domains, such as sport and engineering. Our project will test the effect of CI on the long-term retention of BLS skills. We hypothesize that participants trained in BLS using CI techniques will have superior skill retention at 3 months compared to those trained with the conventional BLS course.

DETAILED DESCRIPTION:
Current BLS courses deliver a curriculum in which learners go through several basic stations in a sequence organized by the American Heart Association (AHA). Learners spend a fixed amount of time at each station, once, thus switching task as many times as the number of stations. This blocked practice design is easy to implement and manage and could also be a contributing factor to the poor retention of BLS skills in laypeople (11). In the next three paragraphs, we highlight why contextual interference is beneficial for skill retention, how contextual interference can be beneficial for medical skills training and why the benefits of contextual interference are particularly relevant for BLS training.

Contextual interference (CI) is a practice scheduling method that involves presenting skills (or stations) in a sequential or random order. Each skill or station is presented multiple times during a learning session (i.e., performing for a shorter duration at each station, but returning multiple times). Both random and sequential order schedules can yield comparable learning benefits (19). With a CI practice schedule, skills are partially forgotten while learners are practicing other skills. As a result, the learner must actively recall each skill multiple times. These repeated memory retrieval processes facilitate better retention after CI practice, compared to a blocked practice schedule (19). A simple analogy can be made with learning multiplication tables: once one has tried 7 times 9, the exercise is not as beneficial for learning if one tried 7 times 9 again on the next trial. Having to retrieve information multiple times with other skills (or time) between trials maximizes long-term skill retention (19). CI is also beneficial when practiced skills are distinct from each other (12). Because many skills are being processed at the same time, the learner must create distinctive memories for each skill. Altogether, the repeated recalls and contrasts involved in CI may have a negative effect on immediate performance (i.e. immediate testing), but typically have a positive effect on long-term learning (i.e. retention) (13). More relevant to this project, the positive effects of CI extend from the motor to the verbal-cognitive domain and have been replicated with various skills levels and learner age groups (14).

Contextual interference has been shown to improve long-term learning among engineers in training of troubleshooting skills (15). Although well studied in sport and other areas outside healthcare, CI has been less well studied in medical education with only a few studies on surgical procedural tasks. Not all implementations of contextual interference have yielded better skill retention and transfer compared to blocked practice (16, 17). In this project, contextual interference will be carefully tested for BLS training by optimizing subtask transitions. In surgical procedures, for instance, CI studies have involved breaking a complex sequential task or procedure into subtasks and implementing CI practice with arbitrarily organized subtasks. An issue with that approach is that learners miss the opportunity to practice the transition from one subtask to another, which can hinder learning. Conversely, BLS skills stations are distinct from each other, technically simple, and do not require complex transitions between skills.

The last but not least relevant factor is that BLS requires transferring the skill into an unpracticed context (13). While orthopedic surgery is learned and performed in fairly comparable and repeatable conditions, BLS is learned in a classroom but needs to be transferred wherever a cardiac arrest takes place. Because contextual interference not only favours better retention but also better transfer to new situations (20), it is imperative to test if such a practice can lead to better BLS skill retention and transferability than conventional blocked practice schedules.

The proposed study will compare skill retention among a group of laypeople being taught BLS using the current standard teaching program compared to those exposed to a CI based program. We hypothesize that participants trained in BLS using a contextual interference practice schedule will have superior skill retention at a retention post-test, 3 months after training, compared to the standard blocked practice schedule employed in current BLS training sessions. This study will be a single-blinded randomized controlled trial. Ethical approval will be obtained from the Ottawa Health Science Research Ethics Board prior to recruitment. Written informed consent and a confidentiality agreement will be obtained from all participants.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18

Exclusion Criteria:

* Health issues preventing them from performing BLS skills
* Previous BLS training

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2015-07; Primary Completion 2017-04 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Full BLS performance on the retention post-test | 3 months
  Participants will repeat a BLS test at 3 months.

SECONDARY OUTCOMES:
Time to start chest compressions, defibrillation using AED | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada